CLINICAL TRIAL: NCT05912504
Title: Long Term Follow-up of Vertebral Compression Fracture In-patients Treated With Integrated Complementary and Alternative Medicine: A Retrospective Chart Review and Survey
Brief Title: Long Term Follow-up of Vertebral Compression Fracture In-patients Treated: A Retrospective Chart Review and Survey
Status: Completed | Type: Observational
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Other Study IDs: JS-CT-2023-01
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Vertebral Compression Fracture; Korean Traditional Medicine; Integrative Korean Medicine; Vertebral Compression
Keywords: Compression Fracture; Integrated Complementary and Alternative Medicine:
MeSH Terms: conditions — Fractures, Compression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Phoen survey — A questionnaire about the current symptoms and satisfaction for received treatment will be conducted over the phone for patients.

SUMMARY:
The purpose of this study is to reveal the effectiveness and safety of integrative Korean medicine for Vertebral Compression Fracture in-patients by observing inpatients treated with integrative Korean medicine.

This study is a retrospective observational study. The subjects for study are patients diagnosed with Vertebral Compression Fracture and who have been admitted to four Jaseng Hospital of Korean medicine (Gangnam, Bucheon, Daejeon, and Haeundae) for 2016.04.01-2022.06.30.

Medical records of selected patients will be analyzed, and telephone surveys will be conducted for each patient. The survey questions are Numeric ratinc scale (NRS), Oswestry Disability Index(ODI), quality of life, and Patient Global Impression of Change (PGIC), etc.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with Acute Compression Fracture' of thoracic or lumbar vertebrae from EMR X-ray or MRI, CT imaging (The temporal criterion for dividing acute and chronic compression fractures was based on 3 months after symptoms began in the case of compression fractures caused by osteoporosis, and acute and chronic were also divided based on 3 months after trauma.)
2. Patient hospitalized for more than a week
3. Pateints above 19 years old and below 80 years old
4. Patients who have agreed to participate the study

Exclusion Criteria:

1. Where the vertebral fracture is not a vertebral body, but a transverse protrusion, a polar protrusion, etc.
2. Other chronic conditions that may interfere with the interpretation of treatment effects or outcomes: cardiovascular disease, kidney disease, diabetic neuropathy, dementia, epilepsy, etc.
3. If the cause of pain is due to soft tissue disease, not the spine: tumor, fibromyalgia, rheumatoid arthritis, gout, etc.
4. a person with a congenital spinal disorder
5. For patients within 3 months of spinal surgery
6. A person who is unable to communicate normally due to dementia or mild cognitive impairment;
7. Other cases where the researcher is not suitable for participation in the study.
8. Those who do not agree to participate in the study.

Ages: 19 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Recruit people who meet the selection criteria and conduct a telephone survey.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) | [Time Frame: Finish survey by November 2023]
  NRS uses an 11-point scale to evaluate current neck pain and radiating pain where no pain is indicated by '0', and the worst pain imaginable by '10'. NRS was assessed at admission, 2 weeks after admission, discharge, and long term follow up.

SECONDARY OUTCOMES:
Oswestry Disability Index(ODI) | [Time Frame: Finish survey by November 2023]
  ODI is a 10-item questionnaire developed to evaluate the degree of disability for lower back pain. Each item is divided into 6 levels, and 0 to 5 points are awarded. The higher the score, the greater the degree of disability. The investigators will conduct an validated Korean NDI questionnaire
The five level version of EuroQol-5 Dimension (EQ-5D) | [Time Frame: Finish survey by November 2023]
  EQ-5D is most widely used as a method of indirectly calculating the quality of life from various aspects. The EQ-5D-5L consists of 5 questions (mobility, self-care, usual activities, pain, anxiety/depression) that ask about the current state of health, and answers each question with 5 likert. (1=I have no problems about, 2=I have slight problems about, 3=I have moderate problems about, 4=I have severe problems about, 5=I am unable to about) In this study, the validated Korean version questionnaire will be used.
Patient Global Impression of Change (PGIC) | [Time Frame: Finish survey by November 2023]
  PGIC is an indicator that evaluates the improvement of patients in 7 steps, and the subject responds with improvement of functional limitation after treatment with 7 likert. (1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, 7=very much worse).
Spine Operation | [Time Frame: Finish survey by November 2023]
  Operation status
Treatment after discharge survey | [Time Frame: Finish survey by November 2023]
  Treatment history after discharge
Satisfaction with integrative Korean medicine survey | [Time Frame: Finish survey by November 2023]
  Preference for integrative Korean medicine, satisfaction with integrative Korean medicine, How helpful hospitalization has been for returning to work and adjusting to daily life.

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, Dr, Study Chair — Bucheon Jaseng Hospital of Korean Medicine
Locations (1):
- Bucheon Jaseng Hospital of Korean Medicine, Bucheon-si, Gyeonggi Province, South Korea

IPD SHARING:
Plan to Share IPD: No